CLINICAL TRIAL: NCT06596980
Title: Single Arm Study Assessing the Effect of the Digital Medical Device Poppins Clinical for Cognitive and Musical Training in Pediatric Participants With a Specific Learning Disability With Deficits in Reading
Brief Title: Examining the Effect of a Digital Medical Device for Cognitive and Musical Training in Children With Reading Disabilities
Acronym: POPPINS-CE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poppins (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POPPINS-CE; 2024-A00432-45 (Other: ANSM)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Learning Disorders, Specific; Learning Disabilities; Specific Learning Disorder, With Impairment in Reading; Dyslexia
MeSH Terms: conditions — Specific Learning Disorder; Learning Disabilities; Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Use of the medical device Poppins Clinical 5 times per weeks (20 minutes training sessions)
  Interventions: Device: Poppins Clinical

INTERVENTIONS:
Device: Poppins Clinical — Poppins Clinical is a software as a medical device that combines a musical and cognitive training program and written language training program.

SUMMARY:
The goal of this clinical trial is to assess the effect on reading skills of the digital medical device Poppins Clinical for cognitive and musical training in pediatric participants (ages 7-11) with a specific learning disability with reading deficit. The main objective of the study is to assess the evolution in reading skills through a word reading task before and after the intervention.

Participants will be asked to train with the digital medical device Poppins Clinical 5 times per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLD with reading deficit, based on a speech-language assessment. SLD with reading deficit is defined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5-TR, 2022) and the International Classification of Diseases (ICD-11, 2022). The speech-language assessment should consist of at least three reading and/or transcription tests with a SD (standard deviation) of at least - 1.4 or a result below the 20th percentile or two reading and/or transcription tests with a SD of at least - 2 SD or a results below the 10th percentile;
* Subject aged between 7 and 11, enrolled from CE1 to CM2;
* French mother tongue or French bilingualism at home and more than 3 years schooling in France;
* Tablet or smartphone available at home;
* Subject affiliated to the French National Insurance (Securite Sociale)
* Subject and parental/legal guardians consent to participate, and commitment to follow the protocol.

Exclusion Criteria:

* Subject has previously used Poppins Clinical or Mila-Learn;
* Uncontrolled chronic illness (at investigator's discretion);
* Previous epileptic seizures;
* Participant actively participating in an interventional study that may affect results.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Effect of Poppins Clinical on reading abilities (accuracy) | 8 weeks
  Evaluate the effect of 8 weeks of training with Poppins Clinical on reading abilities (in terms of reading accuracy) of participants using a word reading task and measuring the number of correctly read words.

SECONDARY OUTCOMES:
Reported adverse events | 8 weeks
  To evaluate safety, reported adverse events during the 8 weeks follow-up phase will be evaluated.
Effect of Poppins Clinical on reading abilities (speed) | 8 weeks
  Evaluate the effect of 8 weeks of training with Poppins Clinical on reading abilities (in terms of speed) of participants using a word reading task and measuring the number of read words.
Effect of Poppins Clinical on phonological skills | 8 weeks
  Evaluate the effect of 8 weeks of training with Poppins Clinical on phonological skills of participants using the BALE test.
Comparison of the effect of Poppins Clinicals to a former version of the device on reading abilities (accuracy) | 8 weeks
  Compare the effect of Poppins Clinical to the effect of the former version of the medical device (Mila-Learn) on reading abilities (in terms of reading accuracy) using a word reading task and measuring the number of correctly read words.
Comparison of the effect of Poppins Clinicals to a former version of the device on reading abilities (speed) | 8 weeks
  Compare the effect of Poppins Clinical to the effect of the former version of the medical device (Mila-Learn) on reading abilities (in terms of reading speed) using a word reading task and measuring the number of read words.

CONTACTS AND LOCATIONS:
Overall Officials: David Cohen, Principal Investigator — Hôpital Pitié-Salpêtrière, Paris, France
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grossard C, Descamps M, Pellerin H, Vonthron F, Cohen D. Children's Improvement After Language and Rhythm Training With the Digital Medical Device Poppins for Dyslexia: Single-Arm Intervention Study. JMIR Serious Games. 2025 Aug 1;13:e76435. doi: 10.2196/76435. PMID 40750096